CLINICAL TRIAL: NCT03988218
Title: Perception and Representation of Internal Body in Anorexia Nervosa
Acronym: PERCEPCOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Aude Paquet, PhD, Centre Hospitalier Esquirol
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: percepcor
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Anorexia Nervosa
Keywords: Body awareness; Interoceptive awareness; Anorexia Nervosa; Adolescent; Body image
MeSH Terms: conditions — Anorexia Nervosa | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anorexia (Experimental): Subjects with anorexia nervosa
  Interventions: Behavioral: perceptive tests
- Control (Active Comparator): Subjects without eating disorders
  Interventions: Behavioral: perceptive tests

INTERVENTIONS:
Behavioral: perceptive tests — many tests are realized: a drawing of the interior of the body a heartbeat detection test an ischemia induction test many scales: Eating Attitude Test; Body Awareness Questionnaire; Body Shape Questionnaire; Hospital Anxiety and Depression; Questionnaire de Satisfaction Corporelle et de Perception Globale de Soi
  Other Names: scales

SUMMARY:
This study focuses on representations of the interior of the body and interoceptive awareness in women with anorexia nervosa in comparison with women without eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa according to DSM-5
* aged above than 14
* BMI between 14 and 18.5 for adults or less than the reference age by age for minors

Exclusion Criteria:

* Unable to understand the tests, poor understanding of the French language
* Mental retardation
* Severe psychiatric comorbidity (bipolar disorder, schizophrenia)
* Lesion or pathology of the upper limbs
* Pregnancy
* Absence of social protection
* Hospitalization under duress

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
drawing | At inclusion
  Number and nature of organs drawn

SECONDARY OUTCOMES:
IAI | At inclusion
  interoceptive awareness index
Time | At inclusion
  time to obtain a score of 3 on the analogue visual scale at the ischemia induction test

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Esquirol, Limoges, France

REFERENCES:
- [Derived] Paquet A, Girard M, Passerieux C, Boule MC, Lacroix A, Sazerat P, Olliac B, Nubukpo P. The body interior in anorexia nervosa: from interoception to conceptual representation of body interior. Front Psychol. 2024 Jun 24;15:1389463. doi: 10.3389/fpsyg.2024.1389463. eCollection 2024. PMID 38979073